CLINICAL TRIAL: NCT06467773
Title: An Oberservational Study of Utility of TSPO-PET/MRI Using the Radiotracer ([18F]-DPA-714) in Surveillance of Neuroinflammation in the Central Nervous System
Brief Title: TSPO-PET/MRI in Surveillance of Neuroinflammation in the Central Nervous System
Status: Recruiting | Type: Observational
Sponsor: Tongji Hospital (Other)
Collaborators: Jianmin Pharmaceutical Group Co., LTD. (Industry)
Responsible Party: Principal Investigator, Wei Wang, Professor of Neurology, President of Tongji Hospita, Tongji Hospital
Other Study IDs: PETinCNS
Record Dates: First submitted 2024-06-12; First posted 2024-06-21 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Central Nervous System Diseases
MeSH Terms: conditions — Central Nervous System Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, cerebrospinal fluid or feces
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ICVD: ischemic cerebrovascular diseases
  Interventions: Radiation: Radiation: PET-MRI with [18F]-DPA-714
- Neurological Autoimmune Diseases: Multiple Sclerosis，Neuromyelitis Optica Spectrum Disorders and Autoimmune Encephalitis
  Interventions: Radiation: Radiation: PET-MRI with [18F]-DPA-714
- other: other encephalomyelitis
  Interventions: Radiation: Radiation: PET-MRI with [18F]-DPA-714

INTERVENTIONS:
Radiation: Radiation: PET-MRI with [18F]-DPA-714 — Radiation: PET-MRI with [18F]-DPA-714

SUMMARY:
Central Nervous System (CNS) inflammation is an immune response activated in the brain and spinal cord by microglial cells and astrocytes, commonly occurring under conditions such as central nervous system ischemia, autoimmunity, infection, toxins, and trauma.

Microglial cells, as the innate immune cells of the central nervous system, are responsible for driving the inflammatory response and play a crucial role in sensing environmental changes, responding to harmful stimuli, and engulfing dead neurons. They also present antigens to T lymphocytes, mediating interactions between the peripheral immune system and the central nervous system. Factors released by neuronal cells can either promote or inhibit inflammation, and monitoring the level of inflammation driven by microglial cells is essential for the diagnosis and treatment of central nervous system diseases.

MRI is the primary imaging method for central nervous system inflammation, but it can be challenging to diagnose. PET/MR, a technology that integrates PET and MR imaging, provides high-quality diagnostic images and is valuable for the early detection, diagnosis, and assessment of central nervous system diseases. The radioactive ligand 18F-DPA-714 PET, targeting the translocation protein (TSPO), can visualize activated microglial cells, which may have a gain effect in detecting active central nervous system inflammation.

This study aims to explore the application of 18F-DPA-714 PET/MR in the early diagnosis, treatment evaluation, and prognosis of central nervous system inflammation.

ELIGIBILITY:
Inclusion Criteria:

-Clinical diagnosis of ischemic stroke, autoimmune ecephalitis, Neuromyelitis optica spectrum disorders, or multiple sclerosis, etc.al

Exclusion Criteria:

* Claustrophobia
* Metal Implants
* Pregancy
* Breast-feeding
* Renal insufficiency (GFR < 60 mL/min/1.73m2)
* Allergy or other contraindication to gadolinium-based MR contrast agent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients diagnosis with central nervous system diseases (lesions occurring in the brain or spinal cord, such as stroke, autoimmune encephalitis, neuromyelitis optica spectrum disorders, multiple sclerosis, etc.)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2029-06 (Estimated); Study Completion 2029-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in TSPO Radiotracer Uptake | 12 months
  Quantify the regional neuroinflammatory load, measured as binding of PET tracer to TSPO.

SECONDARY OUTCOMES:
Free Diffusing Water Fraction | 12 months
  Calculated using MR-DWI
Peripheral Levels of Pro-Inflammatory Cytokines | 12 months
  Evaluated using blood samples, including IL-6, IL-4, IL-10, hs-CRP and PCT etc,al
CSF Levels of Pro-Inflammatory Cytokines | 12 months
  Evaluated using cerebrospinal fluid, IL-6, IL-4, IL-10, hs-CRP and PCT etc, al
CSF Levels of neural injury markers | 12 months
  Evaluated using cerebrospinal fluid, GFAP, NFL and sTREM2 etc, al
MRI Correlation | 12 months
  Correlation of white matter lesion volume and MRI measures of white matter tract injury determined from DTI with measures of TSPO uptake
Inflammatory Markers correlation | 12 months
  Correlation of PET derived measures of TSPO uptake with inflammatory markers (IL-6, IL-4, IL-10, hs-CRP and PCT etc, al) in the blood or cerebrospinal fluid
Neural injury markers correlation | 12 months
  Correlation of PET derived measures of TSPO uptake with neural injury markers ( GFAP, NFL and sTREM2) in the cerebrospinal fluid

CONTACTS AND LOCATIONS:
Overall Officials: Wei Wang, MD, Principal Investigator — Tongji Hospital
Locations (1):
- Tongji Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Shi K, Tian DC, Li ZG, Ducruet AF, Lawton MT, Shi FD. Global brain inflammation in stroke. Lancet Neurol. 2019 Nov;18(11):1058-1066. doi: 10.1016/S1474-4422(19)30078-X. Epub 2019 Jul 8. PMID 31296369
- [Result] Kwon HS, Koh SH. Neuroinflammation in neurodegenerative disorders: the roles of microglia and astrocytes. Transl Neurodegener. 2020 Nov 26;9(1):42. doi: 10.1186/s40035-020-00221-2. PMID 33239064
- [Result] Voet S, Prinz M, van Loo G. Microglia in Central Nervous System Inflammation and Multiple Sclerosis Pathology. Trends Mol Med. 2019 Feb;25(2):112-123. doi: 10.1016/j.molmed.2018.11.005. Epub 2018 Dec 18. PMID 30578090
- [Result] Kreisl WC, Kim MJ, Coughlin JM, Henter ID, Owen DR, Innis RB. PET imaging of neuroinflammation in neurological disorders. Lancet Neurol. 2020 Nov;19(11):940-950. doi: 10.1016/S1474-4422(20)30346-X. PMID 33098803
- [Result] Zhang M, Meng H, Zhou Q, Chunyu H, He L, Meng H, Wang H, Wang Y, Sun C, Xi Y, Hai W, Huang Q, Li B, Chen S. Microglial Activation Imaging Using 18F-DPA-714 PET/MRI for Detecting Autoimmune Encephalitis. Radiology. 2024 Mar;310(3):e230397. doi: 10.1148/radiol.230397. PMID 38441089